CLINICAL TRIAL: NCT01881802
Title: Study of Opioid Immunosuppressive Effects
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaohong Long, doctoral candidate, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 01
Record Dates: First submitted 2013-06-03; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Opioid Abuse or Dependence
Keywords: Opioid drug Abuse; Morphine; Immune Function
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The refrigerator - 80 degrees
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- morphine or heroin dependence patients
- normal control group

SUMMARY:
This trial aims to investigate the effects of opioid-inducing immune suppression on opioid drug abused patients. The methods of the investigators research mainly includes the expression of morphine-related miRNAs in peripheral blood mononuclear cells and cytokine in plasma.

ELIGIBILITY:
Inclusion Criteria:

* subjects were excluded if they had a chronic systemic illness (cardiac, renal, pulmonary, hepatic, endocrine, metabolic, or autoimmune disorders) or
* a major psychiatric disorder or
* if they were abusing substances other than heroin (as determined by urine drug test result). For women, pregnancy was also a reason for exclusion.

Exclusion Criteria:

* Control subjects with no history of drug or alcohol abuse were also excluded if they had
* major medical or psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Guangzhou Psychiatric Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
real-time quantitative polymerase chain reaction | up to 2 months

SECONDARY OUTCOMES:
enzyme-linked immuno sorbent assay | up to 2 months